CLINICAL TRIAL: NCT06749041
Title: Clozapine OpTimal Timing for Optimal moNitoring and Side Effects
Brief Title: Nor)Clozapine Kinetics and Side Effects in Therapy Resistant Schizophrenia and the Optimal Sampling Time for Therapeutic Drug Monitoring
Acronym: COTTONS
Status: Not yet recruiting | Type: Observational
Sponsor: GGZ Noord-Holland-Noord (Other)
Responsible Party: Sponsor
Other Study IDs: COTTONS-v2-22/11/2024
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Side Effects of Clozapine; Neutropenia Due to Clozapine; General Side Effects of Clozapine; Constipation Due to Clozapine; Symptoms of Schizophrenia; Optimal Blood Sampling Time for Clozapine in Patients Who Receive Clozapine Once and Twice Daily; Clozapine and Norclozapine Plasma Level Concentrations
Keywords: cardiovascular side effects; neutropenia; general side effects of clozapine; constipation; symptoms of schizophrenia; optimal blood sampling time; clozapine and norclozapine plasma level concentrations
MeSH Terms: conditions — Neutropenia; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Clozapine and norclozapine concentrations, fasting glucose, serum level HbA1c, insulin, HOMA-IR, triglycerides, HDL, LDL, total cholesterol, the absolute neutrophil count (ANC), inflammation markers, phenylalanine and tyrosine, the genes CYP2C19 and CYP3A4 and genes related to metabolic markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with treatment resistant schizophrenia spectrum disorders receiving clozapine.: Adult patients (age between 18 and 70) with treatment resistant schizophrenia of schizoaffective disorder, treated with oral, once or twice-daily clozapine.

SUMMARY:
The goal of this observational study is to better understand how clozapine treatment can be tailored as regards minimizing side effects and optimizing efficacy and monitoring. Firstly, how clozapine is broken down into norclozapine in the liver and how both clozapine and norclozapine affect side effects are examined. In order to investigate this metabolization process in the liver inflammation levels in the blood are assessed, which inhibit the conversion of clozapine into norclozapine. In addition, various factors related to physical health are assessed, such as blood sugar, cholesterol, weight, waist circumference, blood pressure and heart rate. The role of hormones is investigated, such as cortisol, a stress hormone that affects metabolism and stress levels. Amino acids are examined, which are building blocks of proteins, and specific parts of DNA that influence clozapine metabolism. In addition, investigation follows whether 12 hours after ingestion is a well-chosen time at which the amount of clozapine is measured in the blood in case of ingestion once a day and twice a day. Finally, specific side effects of clozapine are assessed - with special attention to stool - and the severity of the psychiatric symptoms in patients with therapy resistant schizophrenia spectrum disorders.

DETAILED DESCRIPTION:
Rationale:

Therapeutic drug monitoring (TDM) is essential for clozapine and can enhance therapeutic outcomes and minimize side effects. As of yet, research on (nor)clozapine concentrations and their association to metabolic side effects is limited and inconclusive. Unfortunately, not enough is known about individual risk factors for developing metabolic side effects to personalize clozapine treatment. It would be desirable to have another way to predict which clozapine users are at increased risk of developing severe side effects. Current guidelines are based on limited evidence, potentially resulting in inconsistent or suboptimal monitoring and management.

Objective:

The primary objective is to evaluate the correlation between (nor)clozapine kinetics and serum level HbA1c. Secondary objectives include validating an existing population pharmacokinetic model, assessing the validity of the current 12-hour post-intake sampling practice, determining the optimal sampling window for once-daily clozapine TDM and assessing the correlation of other metabolic and multiple laboratory parameters and influence of demographic and clinical parameters on the pharmacokinetics and -dynamics of clozapine and norclozapine.

ELIGIBILITY:
Inclusion Criteria:

* Standard treatment of a stable, oral dose of clozapine for at least one week (at steady state).
* Age between 18-70 years.
* Registered time of intake as well as sampling time and dosage.
* Registered smoking status (yes/no).
* At least two samples in the elimination phase of clozapine with both clozapine and norclozapine measured.
* Measurement of the white cell count at least every three months or more often.
* Routine metabolic screening performed at moment of inclusion.
* Subjects should be able to understand the study information and procedures and give informed consent or when incapacitated subjects are not reliably able to give informed consent their legal representatives should give informed consent under the condition that these subjects are willing to participate.

Exclusion Criteria:

* Pregnancy.
* Malignancy or treatment with immunosuppressive medication.
* Samples where cessation, start or dose change of interacting co-medication (such as valproic acid, gemfibrozil, fluvoxamine, omeprazole and cyclic oral contraceptives [21 on, 7 days off]) or changes in use of tobacco containing products occurred within seven days prior to blood sampling (21, 28, 34, 35).
* Acute inflammation, infection or samples shortly after intoxication. In case this information is unknown, it may be derived by large unexpected change in levels compared to previous or target levels.
* Not sampled at Starlet (blood collection site) or sampled by dried blood spot
* Unknown status of smoking (including vaping).
* Unknown time of intake of clozapine.
* Unknown time of blood sampling.
* If informed consent is not obtained by the patient or by a legal representative in a mentally incapacitated patient, i.e. a legally incompetent adult.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes adult patients (age between 18 and 70) with treatment resistant schizophrenia of schizoaffective disorder, treated with oral, once or twice-daily clozapine. Data will be collected from mental healthcare organization GGZ-NHN. All the patients have been treated with clozapine as part of standard care, as well as sampled routinely as part of standard care.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-23 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum level HbA1c and (nor)clozapine concentrations and ratio. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  Assessed using a PK-PD turn over model.

SECONDARY OUTCOMES:
Validation of an existing population pharmacokinetic model, assessing the validity of the current 12-hour post-intake sampling practice, determining the optimal sampling window for once-daily clozapine TDM. | For the secondary endpoint pertaining to the sample times retrospective data will be collected from 01-02-2024 up to 01-02-2025.
  The predictive performance of the model by Beex et al. (2023) for our population will be assessed through calculations of the prediction error for each observation as well as the root mean square error to measure the overall prediction accuracy.
  2. Percentage difference in clozapine and norclozapine median concentrations predicted 10, 11, 13 and 14-hour post intake (based on clinical samples) compared to median concentrations at current reference sampling time of 12-hour post intake.
  3. Percentage difference in clozapine and norclozapine concentrations based on different sampling times across entire concentration-time profiles to identify optimal sampling time or window within current therapeutic window of 350-700 μg/L.
The validity of the current 12-hour post-intake sampling practice. | For the secondary endpoint pertaining to the sample times retrospective data will be collected from 01-02-2024 up to 01-02-2025.
  Percentage difference in clozapine and norclozapine median concentrations predicted 10, 11, 13 and 14-hour post intake (based on clinical samples) compared to median concentrations at current reference sampling time of 12-hour post intake.
The optimal sampling window for once-daily clozapine therapeutic drug monitoring. | For the secondary endpoint pertaining to the sample times retrospective data will be collected from 01-02-2024 up to 01-02-2025.
  Percentage difference in clozapine and norclozapine concentrations based on different sampling times across entire concentration-time profiles to identify optimal sampling time or window within current therapeutic window of 350-700 μg/L.
The influence of demographic and clinical parameters on the pharmacokinetics and -dynamics of clozapine and norclozapine. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  Effect of covariates on the pharmacokinetics of clozapine, the metabolite norclozapine (and clozapine/norclozapine ratio). Covariates to be studied include: age, estradiol, comedication (e.g. fluvoxamine), ethnicity, pharmacogenetics, smoking behaviour, inflammation markers, phenylalanine and tyrosine.
The correlation of other metabolic and multiple laboratory parameters on the pharmacokinetics and -dynamics of clozapine and norclozapine. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  Correlation between other metabolic parameters (such as fasting glucose, insulin, HOMA-IR, triglycerides, HDL, LDL, total cholesterol, BMI, abdominal circumference, blood pressure and heart rate)..
Correlation between absolute neutrophilic count (ANC) and total white cell count (WCC) and the (nor)clozapine concentrations and ratio. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  Correlation between ANC and TWC and the (nor)clozapine concentrations and ratio will be assessed using a PK-PD turn over model.
Correlation between general side effects of clozapine and the (nor)clozapine concentrations and ratio. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  Correlation between Glasgow Antipsychotic Side-effect Scale (GASS-C) and the (nor)clozapine concentrations and ratio will be assessed using a PK-PD turn over model.
Correlation between constipation and the (nor)clozapine concentrations and ratio. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  Correlation between the Bristol Stool Form Scale (BSFS) and the (nor)clozapine concentrations and ratio will be assessed using a PK-PD turn over model.
Correlation between symptoms of schizophrenia and the (nor)clozapine concentrations and ratio. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  Correlation between the Positive and Negative Syndrome Scale (PANSS-6) and the (nor)clozapine concentrations and ratio will be assessed using a PK-PD turn over model.
The effect of cortisol concentration and genetics on the correlation of (nor)clozapine concentrations and/or ratio on the metabolic markers. | For each patient two years of follow-up will be collected (until a maximum of 01-12-2027).
  The influence of cortisol concentration and genetics on (nor)clozapine concentrations and/or ratio on the metabolic markers.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bank, PharmD, PhD, Principal Investigator — North West Clinics

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT06749041/Prot_SAP_001.pdf